CLINICAL TRIAL: NCT00105950
Title: A Phase II Study to Evaluate the Efficacy, Safety and Pharmacodynamics of Lapatinib in Patients With Relapsed or Refractory Inflammatory Breast Cancer
Brief Title: Study Of Lapatinib In Patients With Relapsed Or Refractory Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF103009; NCT00214409 (obsolete NCT alias); NCT00278317 (obsolete NCT alias)
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-05

CONDITIONS: Neoplasms, Breast
Keywords: ErbB2 overexpressing; ErbB1 expressing; relapsed breast cancer; refractory inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib (Experimental): Single arm study of lapatinib with no comparator arm.
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — Tyrosine kinase inhibitor administered daily at 1500 mg/kg

SUMMARY:
This study was designed to determine how effective and safe a new investigational drug, lapatinib, is in treating patients with treatment refractory or relapsed inflammatory breast cancer. Tumor tissue collected pre-treatment and at Day 28 will be examined for biologic activity by IHC (immunohistochemistry). Treatment will consist of daily oral therapy with lapatinib. A patient may continue treatment as long as they are receiving benefit. Blood samples for hematology and chemistry panels, MUGA/ECHO (multigated acquisition/echocardiogram) exams and physical exams will be performed throughout the study to monitor safety.

DETAILED DESCRIPTION:
This Phase II open label, multicenter study is designed to evaluate the efficacy, safety, and pharmacodynamic effects of oral lapatinib administered as a single agent therapy to patients with relapsed or refractory inflammatory breast cancer. Eligible patients must have a diagnosis of inflammatory breast cancer based on clinicopathologic criteria, tumor that is readily accessible for biopsy, and must have previously received treatment with an anthracycline and taxane-containing regimen (30 patients) plus trastuzumab (90 patients). Patients enrolled must have tumors that overexpress ErbB2, with or without co-expression of ErbB1. The primary objective for this study is to evaluate the objective response rate (defined as complete response plus partial response). Secondary objectives are to evaluate clinical benefit including quality of life parameters, progression-free survival, overall survival, time-to-response, response duration, safety and tolerability, pharmacodynamic effects on intracellular mediators that regulate tumor cell growth and survival, as well as effects on proteomic profile, and circulating levels of extracellular domains of ErbB1 and ErbB2 in peripheral blood.

ELIGIBILITY:
Inclusion criteria:

* Must have a life expectancy of at least 12 weeks.
* Has a left ventricular ejection fraction (LVEF) ≥ 50%, or ≥ lower limit of normal for the institution, based on ECHO or MUGA.
* Aspartate and alanine transaminase (AST or ALT) ≤ 3 times the upper limit of the reference range (patients with liver metastases may have AST and ALT ≤ 5 times the upper limit of the reference range and may be enrolled).
* Total bilirubin ≤ 3.0 mg/dL.
* Serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance (CrCl) ≥ 30 mL/min
* Adequate bone marrow function. Hemoglobin ≥ 9 gm/dL. Absolute granulocyte count ≥ 1,500/mm³ (1.5 x 10^9/L). Platelets ≥ 75,000/mm³ (100 x 10^9/L).
* Recovered or stabilized sufficiently from side effects associated with previous chemotherapy, surgery or radiotherapy.
* Provided written informed consent.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2.
* Able to swallow and retain oral medication.
* Male or female, if female:

A female is eligible to enter and participate in the study if she is of:

1. Non-childbearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal); or
2. Childbearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate), has a negative serum pregnancy test at screening, and agrees to one of the following where considered acceptable to the local IRB/IEC: Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm).

Abstinence from sexual intercourse from 2 weeks prior to administration of the investigational product, throughout the active study treatment period, and through the post-treatment follow-up visit (to occur 28 days after last dose of investigational product).

Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject.

Implants of levonorgestrel. Injectable progestogen. Any intrauterine device (IUD) with a documented failure rate of less than 1% per year.

Oral contraceptives (either combined or progestogen only). Barrier methods including diaphragm or condom with a spermicide.

* At least 18 years of age.
* Has either measurable disease by Response Evaluation Criteria in Solid Tumors (RESIST) or clinically evaluable skin disease. Measurable lesions may be in the field of prior adjuvant irradiation; however, there must be at least an 8 week period between the last radiation treatment and the baseline scan documenting disease status for the lesion to be measurable.
* Tumor that is accessible for biopsy.
* Tumor that overexpresses ErbB2 defined as 3+ by IHC or FISH +. The ErbB 2 overexpression must be documented prior to dosing.
* Documented disease progression or relapse following treatment, which must have contained a taxane and anthracycline-containing regimen in the adjuvant or metastatic setting (30 patients) plus trastuzumab (90 patients)
* Histological diagnosis of breast carcinoma with a clinical diagnosis of IBC based on the presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast. Pathologic evidence of dermal lymphatic invasion should be noted but is not required for diagnosis.

Exclusion criteria:

* Is clinically assessed to have inadequate venous access for protocol-related blood draws.
* Has a clinically significant electrocardiogram (ECG) abnormality.
* Has Class II to IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Has physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Is currently receiving oral steroid treatment (inhaled steroids are permitted), or any other medication on the prohibited medications list
* Is currently receiving amiodarone or has received amiodarone in the 6 months prior to screening.
* Has received chemotherapy, immunotherapy, biologic therapy or hormonal therapy within the past 14 days, with the exception of mitomycin C within the past 6 weeks.
* Has received treatment with any investigational drug in the previous 4 weeks.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product. These include other anilinoquinazolines, such as gefitinib [Iressa], erlotinib [Tarceva], or other chemically related compounds.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
* Has evidence of symptomatic or uncontrolled brain metastases or leptomeningeal disease. Patients with brain metastases treated by surgery and/or radiotherapy are eligible if neurologically stable and do not require steroids or anticonvulsants.
* Has malabsorption syndrome, a disease affecting gastrointestinal function, or resection of the stomach or small bowel.
* Is a pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Objective Response rate (complete response plus partial response) | Week 84

SECONDARY OUTCOMES:
Clinical benefit (progression free survival, time to progression, response duration) | week 84
Assessment of clinical benefit, defined as CR or PR for at least 4 weeks, or SD for at least 6 months | week 84
Calculation of progression-free survival, defined as the time between the first dose of investigational product and the first documented sign of disease progression or death. | week 84
Calculation of time-to-response, defined as the time between the first dose of investigational product and the first documented CR or PR. | week 84
Calculation of duration of response, defined as the time from initial documented CR or PR to the first documented sign of disease progression. | week 84
Evaluation of changes in QoL and pain scale measurements collected on Day 1 and every 4 weeks while receiving study treatment. | week 84
Evaluation of adverse events (AEs), changes in laboratory values and echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) results from pre-dose, during dosing and post-dose assessments | week 84
Comparison of the effects of lapatinib on biomarkers that are involved in regulating tumor cell proliferation and survival (e.g., phosphorylated forms of Erk1/2 and Akt, STAT3, S6 Kinase, Bad, truncated ErbB2 and potentially other downstream mediators of | Day 28
tumor cell growth and survival) by quantitative IHC and by direct and genome-wide methods (e.g., direct sequencing and DNA microarray) in tumor tissue collected prior to and following 28 days of lapatinib monotherapy. | Day 28
Examination of the effects of lapatinib therapy on the levels of circulating ErbB1 and ErbB2 ECD and the proteomic profile of peripheral blood. Investigation of the use of FDG-PET to predict early response to treatment with lapatinib. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (8):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Zion, Illinois
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Toronto, Ontario, Canada
- France (5):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
- Israel (2):
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Zrifin
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
- Tunisia (2):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Tunis
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Result] Kaufman B, Trudeau M, Awada A, Blackwell K, Bachelot T, Salazar V, DeSilvio M, Westlund R, Zaks T, Spector N, Johnston S. Lapatinib monotherapy in patients with HER2-overexpressing relapsed or refractory inflammatory breast cancer: final results and survival of the expanded HER2+ cohort in EGF103009, a phase II study. Lancet Oncol. 2009 Jun;10(6):581-8. doi: 10.1016/S1470-2045(09)70087-7. Epub 2009 Apr 24. PMID 19394894
- [Result] Kaufman B, Wu Y, Amonkar MM, Sherrill B, Bachelot T, Salazar V, Viens P, Johnston S. Impact of lapatinib monotherapy on QOL and pain symptoms in patients with HER2+ relapsed or refractory inflammatory breast cancer. Curr Med Res Opin. 2010 May;26(5):1065-73. doi: 10.1185/03007991003680323. PMID 20214527